CLINICAL TRIAL: NCT04717245
Title: Comparative Study : The Effect of Vaginal Estrogen Use, Fractional CO2 LASER and Microablative Fractional Radiofrequency in the Treatment of Vaginal Atrophy: Clinical, Histological, Immunohistochemical and Molecular Biology Study
Brief Title: Comparative Study: Vaginal Promestriene Use, Fractional CO2 LASER and Radiofrequency in the Vaginal Atrophy Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAI
Record Dates: First submitted 2018-08-28; First posted 2021-01-22 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2018-08

CONDITIONS: Vaginal Atrophy
Keywords: genital atrophy; fractional CO2 laser; microablative fractional radiofrequency; quality of life; sexuality; promestriene; Menopause genitourinary syndrome
MeSH Terms: conditions — Sexuality | interventions — promestriene

STUDY DESIGN:
Intervention Model Description: In this study, 75 patients were included, divided into these three groups:
  Group 1 - Treatment with topical vaginal promestriene - 25 patients were included in this group
  Group 2 - Treatment with fractional CO2 LASER - 25 patients were included in this group
  Group 3 - Treatment with microablative fractional radiofrequency - 25 patients were included in this group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fractional CO2 LASER (Active Comparator): Vaginal fractional CO2 LASER 3 sessions applications
  Interventions: Other: Fractional CO2 LASER
- Microablative fractional radiofrequency (Active Comparator): Vaginal Microablative fractional radiofrequency 3 sessions application
  Interventions: Other: Microablative Fractional radiofrequency
- Promestriene Vaginal (Active Comparator): Promestriene vaginal use during 3 months
  Interventions: Drug: Promestriene Vaginal

INTERVENTIONS:
Drug: Promestriene Vaginal — Patients used promestriene vaginal cream for 3 months. The use was recommended to be diary fot the first 2 weeks, and then, repeat every 3 days.
  Other Names: Promestrieno
  Arms: Promestriene Vaginal
Other: Fractional CO2 LASER — LASER treatment with fractional CO2 Laser was performed in 3 sessions with intervals of 4 weeks between them. Before each session, the patients underwent specular examination.
  Fractional CO2 LASER was applied following these parameters, fixed in all sessions: vagina wall - power40 W, dwel time 1000 mcs, spacing 1000 mcm and stack 2, vestibule - power 10W, dwel time 500mcs, spacing 300mcg and satck 1
  Arms: Fractional CO2 LASER
Other: Microablative Fractional radiofrequency — Microablative fractional radiofrequency was performed with the equipment calibrated in FRAXX mode, 45W, Low Energy program 40 milliseconds in the vaginal and introitus wall. Lidocaine spray was applied to vaginal introitus before the procedure.
  The patient was in the gynecological position. The vaginal speculum was placed and, afterwards, the vaginal antisepsis was performed with aqueous chlorhexidine and cleaning with 0.9% saline solution.
  All liquid contents were wiped off before beginning the procedure. The fractured tip will be pressed lightly and as perpendicular as possible into the vulvar or vaginal surface, ensuring full contact of all points in the tissue, starting at the lateral vaginal walls and from the proximal to the distal third.
  Arms: Microablative fractional radiofrequency

SUMMARY:
Postmenopausal hypoestrogenism may determine genital atrophy, which may be accompanied by a non-specific inflammatory process and may hinder or even prevent sexual intercourse. In more severe cases, the patient may have local pain that interferes with their daily activities. The best treatment for increasing genital trophism is still estrogen. However, there are women who can not use this therapy or do not want it. Therefore, there is a need for alternatives, such as ablation techniques: use of CO2 LASER and fractional radiofrequency.

The study was carried out at the outpatient clinic of Lower Genital Tract ambulatory of the Discipline of Gynecology, Department of Obstetrics and Gynecology, Clinical Hospital, Faculty of Medicine, University of São Paulo, involving 75 women who were divided after randomization in three groups:

Group 1 - treatment with topical vaginal promestriene (n = 25 patients); Group 2 - treatment with fractional CO2 LASER (n = 25 patients); Group 3 - fractional microablative radiofrequency treatment (n = 25 patients).

An evaluation of the complaints were be performed through questionnaires on sexuality, quality of life and urinary incontinence, as well as biopsies of the vaginal wall for histomorphometric, immunohistochemical and molecular biology study before and after six months of treatment. The duration of the study were fifteen months.

DETAILED DESCRIPTION:
After completing the eligibility criteria, patients signed the consent inform.

Division of groups:

Were included in the study 75 patients, divided into three groups:

Group 1 - Treatment with topical vaginal promestriene - 25 patients in this group were included patients free of systemic or topical hormonal treatment for at 3 months

Group 2 - Treatment with CO2 LASER - 25 patients, in this group were included patients free of systemic or topical hormonal treatment for at 3 months.

Group 3 - Treatment with microablative fractionated radiofrequency - 25 patients in this group were included patients free of systemic or topical hormonal treatment for at least 3 months.

The present study was open and randomized. The randomization was be performed through the software "Test Generator Software Standard Edition"

At the first visit, all patients responded to the clinical questionnaire of female sex quotient (QS-F), the quality of life questionnaire (SF-36) and the urinary incontinence questionnaire.

All patients were submitted to specular gynecological examination to collect cervical-vaginal cytology, biopsy of 1/3 proximal vaginal wall for histological analysis and immunohistochemistry.

After the results of the examinations and possible treatments required, the patients were referred for the proposed treatments according to their randomized group.

Sampling Cytology :Cervical and vaginal oncology cytology were collected through a smear on a slide with fixative.

The histological expression of the following immunohistochemical parameters will be evaluated:

* Presence and density of estrogen receptors
* Vascular density
* Thickness of the epithelium
* Density of collagen fibers
* Vaginal microbiota
* Vaginal pH

In this study, it will be done a Morphological Analysis, a Histomorphometric analysis and e Immunohistochemical analysis.

ELIGIBILITY:
Inclusion Criteria:

Age equal or superior to 40 years and under 65 years

* Clinical menopause - last menstrual period from 1 to 5 years from the date of recruitment
* FSH measurement> 25 IU / ml, estrogen <20 æg / ml
* Patients with vaginal atrophy and clinical and / or sexual symptoms
* Patients without hormonal treatment for at least five years

Exclusion Criteria:

* Whole Hymen

  * Altered oncology cytology of the cervix and / or vagina
  * Vaginal infections
  * Connective tissue diseases
  * Immunosuppression
  * Coagulation change
  * Diabetes Mellitus
  * Thyroid diseases
  * Use of systemic or local feminine hormones
  * Use of other substances with estrogenic properties

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Life's quality questionnaire | 3-4 months
  It was acessed at the beginnig and in the end of the treatment. We used the Short Form Health Survey 36 questionnaire for this parameter. It contains 36 items measuring eight dimensions, that vary the pontuation between 1-5 to 1-6. All but one of the 36 items are used to score the SF-36 eight domains that are aggregated in two summary measures, Physical and Mental components. Among the eight domains, three scales (Physical Functioning, Role-Physical, and Bodily Pain) contributes mostly to the Physical Component Summary (PCS) and three (Mental Health, Role-Emotional, and Social Functioning) contributes to the Mental Component Summary. The domains Vitality, General Health, and Social Functioning present noteworthy correlations with both summary componentNormalized scores below 50 are interpreted as below the generals population. The better is to have a higher pontuation.

SECONDARY OUTCOMES:
Sexuality questionnaire - Female Sexual Function Index | 3-4 months
  This questionnaire analyses 6 parameters: desire, excitation, lubrication, orgasm, satisfaction and pain. Tha maximum pontuation for each parameter is 6, and for the entire questionnaire is 36 (the best pontuation).
pH values | 3-4 months
  We used a pH tape to determine the vaginal pH. The normal measure é between 3,8 and 4,5.
score symptoms | 3-4 months
  Patients describe these symptoms dryness, itching, burnig and pain as absent (0 points); mild :1 point; moderate : 2 points and severe : 3 points, at the begging and in the end of the treatment. The best pontuation is zero and the worst is 12.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Maria Soares Junior, PHD, Study Director — Universidade de São Paulo departamento de ginecologia
Locations (1):
- Disciplina de ginecologia - departamento de ginecologia e obstetrícia - faculdade de medicina da USP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seganfredo IB, Bianchi C, Tacla M, Chedraui P, Haddad JM, Simoes R, Baracat EC, Soares JM Jr. Comparison of promestriene with vaginal fractional CO2 laser and radiofrequency treatments of genitourinary syndrome of menopause. Maturitas. 2024 Aug;186:108008. doi: 10.1016/j.maturitas.2024.108008. Epub 2024 Apr 24. PMID 38714422